CLINICAL TRIAL: NCT01741246
Title: Neuroimaging Studies of Chronic Primary Headaches Using Positron Emission Tomography and Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 1107004
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Migraine; Chronic Migraine
Keywords: Episodic migraine; Chronic migraine; Magnetic resonance imaging; Positron emission tomography
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Headache-free subjects.
- Episodic migraine: Patients with less that 15 headache days per month that fulfill International Classification of Headache Disorders 2R (ICHD-2nd edition Revised)- criteria for Episodic Migraine.
- Chronic migraine: Patients that fulfill International Classification of Headache Disorders (ICHD)-2R criteria for chronic migraine (more than 15 days per month).

SUMMARY:
Investigators hypothesize that chronic primary headaches are accompanied by a discrete pattern of brain metabolism and activity involving brain structures related to the development of acute exacerbations as well as pain modulation. Such structures include the brainstem, hypothalamus, and orbitofrontal cortex and can be defined using functional brain imaging.

DETAILED DESCRIPTION:
Specific aims of the study include:

1. To determine the pattern of brain metabolism using positron emission tomography (PET) found in chronic migraine, episodic migraine and control patients.
2. To determine changes of resting state brain networks using magnetic resonance imaging (MRI) between patients with chronic or episodic headache and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65

  * No medical contraindication.

Chronic headache group:

* Patients with chronic primary headaches who are experiencing phases with background pain as well as habitual pain exacerbations.
* Able to provide informed consent.
* Not pregnant or planning to become so, with a pregnancy test prior to scanning.

Control group and Episodic migraine group:

* Patients with episodic migraine
* Able to provide informed consent.
* Not pregnant or planning to become so, with a pregnancy test prior to scanning.

Exclusion Criteria:

* Taking a migraine preventive currently or in the last fifteen days.
* Known claustrophobia
* Patient is pregnant, planning to be pregnant, or becomes pregnant.
* Patients with metal implants.
* Patients who have had a study involving radiation within the one year prior to enrolling in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with episodic migraine, chronic migraine and control patients. Definitions are taken for the International Classification of Headache Disorders-2nd Edition (see references).
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pattern of brain metabolism using positron emission tomography(PET). | Estimated to be approximately three years post baseline
  Neuroimaging Studies of Chronic Primary Headaches Using Positron Emission Tomography and Magnetic Resonance Imaging to determine the pattern of brain metabolism.
Changes of resting state brain networks using magnetic resonance imaging (MRI) | Estimated to be approximately three years post baseline
  Neuroimaging Studies of Chronic Primary Headaches Using Positron Emission Tomography and Magnetic Resonance Imaging (MRI) To determine any changes of resting state brain networks

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tso, MD, Principal Investigator — University of California, San Francisco; Peter Goadsby, MD PhD, Principal Investigator — University of California, San Francisco; Amy Gelfand, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Background] Welch KM, Goadsby PJ. Chronic daily headache: nosology and pathophysiology. Curr Opin Neurol. 2002 Jun;15(3):287-95. doi: 10.1097/00019052-200206000-00011. PMID 12045727
- [Background] Scher AI, Stewart WF, Liberman J, Lipton RB. Prevalence of frequent headache in a population sample. Headache. 1998 Jul-Aug;38(7):497-506. doi: 10.1046/j.1526-4610.1998.3807497.x. PMID 15613165
- [Background] Bigal ME, Serrano D, Reed M, Lipton RB. Chronic migraine in the population: burden, diagnosis, and satisfaction with treatment. Neurology. 2008 Aug 19;71(8):559-66. doi: 10.1212/01.wnl.0000323925.29520.e7. PMID 18711108
- [Background] Bergerot A, Holland PR, Akerman S, Bartsch T, Ahn AH, MaassenVanDenBrink A, Reuter U, Tassorelli C, Schoenen J, Mitsikostas DD, van den Maagdenberg AM, Goadsby PJ. Animal models of migraine: looking at the component parts of a complex disorder. Eur J Neurosci. 2006 Sep;24(6):1517-34. doi: 10.1111/j.1460-9568.2006.05036.x. PMID 17004916
- [Background] Goadsby PJ, Lipton RB, Ferrari MD. Migraine--current understanding and treatment. N Engl J Med. 2002 Jan 24;346(4):257-70. doi: 10.1056/NEJMra010917. No abstract available. PMID 11807151
- [Background] Afridi SK, Goadsby PJ. Neuroimaging of migraine. Curr Pain Headache Rep. 2006 Jun;10(3):221-4. doi: 10.1007/s11916-006-0049-4. PMID 18778577
- [Background] Weiller C, May A, Limmroth V, Juptner M, Kaube H, Schayck RV, Coenen HH, Diener HC. Brain stem activation in spontaneous human migraine attacks. Nat Med. 1995 Jul;1(7):658-60. doi: 10.1038/nm0795-658. PMID 7585147
- [Background] Bahra A, Matharu MS, Buchel C, Frackowiak RS, Goadsby PJ. Brainstem activation specific to migraine headache. Lancet. 2001 Mar 31;357(9261):1016-7. doi: 10.1016/s0140-6736(00)04250-1. PMID 11293599
- [Background] Afridi SK, Matharu MS, Lee L, Kaube H, Friston KJ, Frackowiak RS, Goadsby PJ. A PET study exploring the laterality of brainstem activation in migraine using glyceryl trinitrate. Brain. 2005 Apr;128(Pt 4):932-9. doi: 10.1093/brain/awh416. Epub 2005 Feb 10. PMID 15705611
- [Background] Afridi SK, Giffin NJ, Kaube H, Friston KJ, Ward NS, Frackowiak RS, Goadsby PJ. A positron emission tomographic study in spontaneous migraine. Arch Neurol. 2005 Aug;62(8):1270-5. doi: 10.1001/archneur.62.8.1270. PMID 16087768
- [Background] Denuelle M, Fabre N, Payoux P, Chollet F, Geraud G. Hypothalamic activation in spontaneous migraine attacks. Headache. 2007 Nov-Dec;47(10):1418-26. doi: 10.1111/j.1526-4610.2007.00776.x. PMID 18052951
- [Background] Goadsby PJ, Hargreaves R. Refractory migraine and chronic migraine: pathophysiological mechanisms. Headache. 2008 Oct;48(9):1399-405. doi: 10.1111/j.1526-4610.2008.01274.x. PMID 19006557
- [Background] Fumal A, Laureys S, Di Clemente L, Boly M, Bohotin V, Vandenheede M, Coppola G, Salmon E, Kupers R, Schoenen J. Orbitofrontal cortex involvement in chronic analgesic-overuse headache evolving from episodic migraine. Brain. 2006 Feb;129(Pt 2):543-50. doi: 10.1093/brain/awh691. Epub 2005 Dec 5. PMID 16330505
- [Background] Valet M, Sprenger T, Boecker H, Willoch F, Rummeny E, Conrad B, Erhard P, Tolle TR. Distraction modulates connectivity of the cingulo-frontal cortex and the midbrain during pain--an fMRI analysis. Pain. 2004 Jun;109(3):399-408. doi: 10.1016/j.pain.2004.02.033. PMID 15157701
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Raichle ME, MacLeod AM, Snyder AZ, Powers WJ, Gusnard DA, Shulman GL. A default mode of brain function. Proc Natl Acad Sci U S A. 2001 Jan 16;98(2):676-82. doi: 10.1073/pnas.98.2.676. PMID 11209064
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Calhoun VD, Adali T, Stevens MC, Kiehl KA, Pekar JJ. Semi-blind ICA of fMRI: A method for utilizing hypothesis-derived time courses in a spatial ICA analysis. Neuroimage. 2005 Apr 1;25(2):527-38. doi: 10.1016/j.neuroimage.2004.12.012. PMID 15784432
- [Background] Matharu MS, Bartsch T, Ward N, Frackowiak RS, Weiner R, Goadsby PJ. Central neuromodulation in chronic migraine patients with suboccipital stimulators: a PET study. Brain. 2004 Jan;127(Pt 1):220-30. doi: 10.1093/brain/awh022. Epub 2003 Nov 7. PMID 14607792
- [Background] Sprenger T, Ruether KV, Boecker H, Valet M, Berthele A, Pfaffenrath V, Woller A, Tolle TR. Altered metabolism in frontal brain circuits in cluster headache. Cephalalgia. 2007 Sep;27(9):1033-42. doi: 10.1111/j.1468-2982.2007.01386.x. Epub 2007 Jul 30. PMID 17666083
- [Background] Headache Classification Committee of The International Headache Society. The International Classification of Headache Disorders (second edition). Cephalalgia 2004;24(Suppl 1):1-160.
- [Background] Frackowiak RS, Friston KJ. Functional neuroanatomy of the human brain: positron emission tomography--a new neuroanatomical technique. J Anat. 1994 Apr;184 ( Pt 2)(Pt 2):211-25. PMID 8014115
- [Background] Talairach J, Tournoux P. Coplanar Stereotaxic Atlas of the Human Brain. New York: Thieme; 1988.
- [Background] Valk PE, Delbeke D, Bailey DL, D.W. T, Maisey MN. Positron Emission Tomography: Springer; 2006.
- [Background] Sprenger T, Seifert CL, Valet M, Staehle KS, Tölle TR, Foerschler A, Zimmer C, Goadsby PJ. Abnormal Interictal Resting State Activity in Episodic Migraine. Presented at the 62nd Annual Meeting of the American Academy of Neurology 2010, Toronto.
- [Background] Headache Classification Committee; Olesen J, Bousser MG, Diener HC, Dodick D, First M, Goadsby PJ, Gobel H, Lainez MJ, Lance JW, Lipton RB, Nappi G, Sakai F, Schoenen J, Silberstein SD, Steiner TJ. New appendix criteria open for a broader concept of chronic migraine. Cephalalgia. 2006 Jun;26(6):742-6. doi: 10.1111/j.1468-2982.2006.01172.x. PMID 16686915